CLINICAL TRIAL: NCT06651060
Title: Comparing the Impact of Climate Labels for Restaurant Menus: a Pilot Study
Brief Title: Climate Labels for Restaurant Menus Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Principal Investigator, Jennifer Falbe, Associate Professor, University of California, Davis
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1641776-8C
Record Dates: First submitted 2024-10-18; First posted 2024-10-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Food Selection
Keywords: Sustainability; Climate change; Diet; Food choices; Food labeling
MeSH Terms: conditions — Food Preferences

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to view a menu based on a real-world restaurant with one of six labeling schemes applied: 1) a QR code on all items (control); 2) High Climate Impact label; 3) High Climate Impact Warning label; 4) Climate Grade label; 5) Climate Grade label also displaying full range of possible grades; 6) Estimated Environmental Cost label. Menus will include main items only. Labels will only appear alongside main menu items and will be assigned using thresholds for greenhouse gas emissions set a priori in kilograms of CO2 equivalent per kilogram of food. Each participant will view a menu based on a real-world restaurant with one of the 6 labels shown on applicable menu items, select the menu item(s) they would like, then respond to survey questions about each label.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Control (QR) labels (Placebo Comparator): Labels placed beneath all menu items will contain QR codes with the text, "scan here", without any mention of sustainability
  Interventions: Behavioral: Menu label
- High Climate Impact labels (Experimental): Labels will be placed beneath menu items with a high climate impact using a predetermined threshold of estimated greenhouse gas emissions set at >=9.2 kgCO2e. Labels will contain white text, "High Climate Impact", on a red background with a globe icon
  Interventions: Behavioral: Menu label
- High Climate Impact Warning labels (Experimental): Labels will be placed beneath menu items with a high climate impact using a predetermined threshold of estimated greenhouse gas emissions set at >=9.2 kgCO2e. Labels will contain white text, "Warning: High Climate Impact", on a red background with a globe icon
  Interventions: Behavioral: Menu label
- Climate Grade labels (Experimental): Labels will be placed beneath all menu items, using predetermined estimated greenhouse gas emission thresholds to assign one of five icon-plus-text labels which indicate a specific climate impact grade (A, B, C, D, and F). Thresholds are set in kgCO2e as follows: [A] <1.7, [B] >=1.7 & <2.6, [C] >=2.6 & <9.2, [D] >=9.2 & <28, [F] >=28. Labels shown will contain white text, "Climate Grade", on a black background with a globe icon. The labels will include a white letter in a colored box on the left side, A (dark green), B (light green), C (yellow), D (orange), or F (red)
  Interventions: Behavioral: Menu label
- Climate Grade label also displaying full range of possible grades (Experimental): Labels will be placed beneath all menu items, using predetermined estimated greenhouse gas emission thresholds to assign one of five icon-plus-text labels which indicate a specific climate impact grade (A, B, C, D, and F). Thresholds are set in kgCO2e as follows: [A] <1.7, [B] >=1.7 & <2.6, [C] >=2.6 & <9.2, [D] >=9.2 & <28, [F] >=28. Labels shown will contain white text, "Climate Grade", on a black background with a globe icon. The labels will include a white letter in a colored box on the left side, A (dark green), B (light green), C (yellow), D (orange), or F (red). This label will also include a small scale of each white letter and colored box option beneath the main white letter and colored box
  Interventions: Behavioral: Menu label
- Estimated Environmental Cost labels (Experimental): Labels will be placed beneath all menu items, displaying the estimated dollar value associated with greenhouse gas emissions. Labels shown will contain white text, "Environmental Cost," with a dollar value (i.e., +$10.90) on a black background with a globe icon
  Interventions: Behavioral: Menu label

INTERVENTIONS:
Behavioral: Menu label — Participants will view a sample of items from a restaurant menu, displayed with labels

SUMMARY:
The aim of this study is to compare responses to 6 different types of labels for restaurant menus: 1) a QR code on all items (control); 2) High Climate Impact label; 3) High Climate Impact Warning label; 4) Climate Grade label; 5) Climate Grade label also displaying full range of possible grades; 6) Estimated Environmental Cost label. Participants will be randomized to 1 of these 6 labeling arms. Each participant will view a menu based on a real-world restaurant with one of the 6 labels shown on applicable menu items, select the menu item they would like, and then respond to survey questions about each label.

DETAILED DESCRIPTION:
This is an online randomized controlled trial in which researchers will use a survey company to recruit participants to an online survey. In the study, participants will be randomized to 1 of 6 labeling arms: 1) a QR code on all items (control); 2) High Climate Impact label; 3) High Climate Impact Warning label; 4) Climate Grade label; 5) Climate Grade label also displaying full range of possible grades; 6) Estimated Environmental Cost label. Labels will only appear alongside main menu items and will be assigned using thresholds for greenhouse gas emissions set a priori in kilograms of CO2 equivalent per kilogram of food. Each participant will view a menu based on a real-world restaurant with one of the 6 labels shown on applicable menu items, select the menu item they would like, then respond to survey questions about each label.

For dichotomous outcomes, the investigators will directly estimate the probability ratio using Poisson regression with a robust error variance, regressing the outcome on indicators for experimental condition. For continuous outcomes, the investigators will use linear regression models, regressing the outcome on indicators for experimental condition. A critical alpha 0.05 will be used, and statistical tests will be two-tailed. Investigators will compare all experimental label conditions to the control label, then compare each experimental label to each other using pairwise comparisons.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* English-speaking
* U.S. residents
* Have eaten restaurant food at least once in the last month
* Participants will reflect the U.S. Census Bureau's American Community Survey estimates for sex, race/ethnicity, educational attainment, and age

Exclusion Criteria:

* Non-US resident
* Younger than 18 years old
* Failing the attention check question
* Completing the survey in less than 33% of the median completion time

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16181 (Actual)
Dates: Start 2024-12-23 (Actual); Primary Completion 2025-02-13 (Actual); Study Completion 2025-02-13 (Actual)

PRIMARY OUTCOMES:
High climate impact menu item selected - dichotomous variable | Up to approx. 1 minutes
  Measured as a dichotomous variable (yes/no) indicating whether participants' hypothetical meal orders include a high climate impact menu item.
Total greenhouse gas emissions - continuous variable | Up to approx. 1 minute
  Cumulative total kilograms of carbon equivalent (kgCO2e) per kilogram of food for all meal items.

SECONDARY OUTCOMES:
Modified Nutrient Profile Index (NPI) score - continuous variable | Up to approx. 1 minute
  NPI scores are based on the UK Ofcom Nutrient Profiling Model, which is used to score individual foods in the U.K. to determine which ones can be marketed to children. The NPI generates a 0 to100-point score for foods and beverages where scores >=64 are considered healthy. NPI scores are based on points awarded from nutrients to encourage (e.g., percent fruits and vegetables, grams of fiber and protein) and nutrients of concern (e.g., sodium, sugar) per 100 grams. For this study, we will generate a modified NPI score to evaluate the healthfulness of full meals comprised of multiple food items. This measure will be determined by calculating the weighted mean NPI score of all food items selected per meal, with each item's NPI score weighted by its proportionate contribution of mass in grams to the total mass of the meal.
  Reference: Rayner, M., Scarborough, P., Boxer, A., & Stockley, L. (2005). Nutrient profiles: development of final model. London: Food Standards Agency.
Total energy (kcal) selected - continuous variable | Up to approx. 1 minute
  The total number of calories in participants' hypothetical meal orders, calculated as the sum of calories across all menu items selected. Higher values indicate more calories selected.
Total saturated fat (g) selected - continuous variable | Up to approx. 1 minute
  The total grams of saturated fat in participants' hypothetical meal orders, calculated as the sum of grams of saturated fat across all menu items selected. Higher values indicate more saturated fat selected.
Total sodium (mg) selected - continuous variable | Up to approx. 1 minute
  The total milligrams of sodium in participants' hypothetical meal orders, calculated as the sum of milligrams of sodium across all menu items selected. Higher values indicate more sodium selected.

OTHER OUTCOMES:
Noticeability - dichotomous variable | Up to approx. 1 minute
  Measured as a dichotomous variable (yes/no) indicating whether participants noticed and can correctly recall the climate, environmental, or control label with the question: "Did you notice any labels (other than calories) next to or below the menu items?." With response options: "Yes, a climate label" (or "Yes, an environmental label" in the environmental cost condition), "Yes, a heart healthy label," "Yes, a vegan label," "Yes, an organic label," "Yes, a local label," "Yes, a QR code label," "No, I did not see a label," "Not sure."
  There is no formal name for this measure. It was developed for this study.
Support - categorical variable | Up to approx. 1 minute
  Measured with a single item: "Imagine the city you live in is considering a policy that would add the label(s) shown below to relevant menu items in chain restaurants. Would you…?" With an image of the assigned label condition the participant was randomized to and the response options: "Strongly oppose this policy," "Somewhat oppose this policy," "No opinion," "Somewhat support this policy," "Strongly support this policy."
  There is no formal name for this measure. It was developed for this study.
Effectiveness - categorical variable | Up to approx. 1 minute
  A single item adapted from the UNC-PME scale to measure how much the climate labels discouraged wanting to purchase an item that has a high climate impact with the question: "How much does this label discourage you from wanting to purchase an item that has a high climate impact?" With response options: "Not at all," "A little bit," "Somewhat," "Quite a bit," and "A great deal."
  Reference: Baig, S. A., Noar, S. M., Gottfredson, N. C., Boynton, M. H., Ribisl, K. M., & Brewer, N. T. (2019). UNC perceived message effectiveness: validation of a brief scale. Annals of Behavioral Medicine, 53(8), 732-742.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Davis, Davis, California, United States

IPD SHARING:
Plan to Share IPD: No